CLINICAL TRIAL: NCT00796744
Title: Randomized, Parallel-Group, Double-Blind, Placebo-Controlled Phase 2 Clinical Trial to Evaluate the Safety and Effectiveness of DSC127 in Treating Subjects With Diabetic Ulcers
Brief Title: Safety and Efficacy Study of DSC127 in Treating Subjects With Diabetic Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Biotest, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DSC127-2008-01
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-08

CONDITIONS: Foot Ulcer, Diabetic; Diabetic Foot
Keywords: Diabetes mellitus; Diabetic neuropathy; Peripheral vascular disease; Infection; Topical application; plantar foot ulcers
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Diabetic Neuropathies; Peripheral Vascular Diseases; Infections | interventions — norLeu3-A(1-7); aclerastide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo Vehicle Control (Placebo Comparator): control placebo vehicle gel
  Interventions: Drug: NorLeu3-A(1-7) in a gel formulation
- 0.03% DSC127 (Active Comparator): 0.03 % DSC127 in Vehicle Control
  Interventions: Drug: NorLeu3-A(1-7) in a gel formulation
- 0.01% DSC127 (Active Comparator): 0.01% DSC127 in Vehicle Control
  Interventions: Drug: NorLeu3-A(1-7) in a gel formulation

INTERVENTIONS:
Drug: NorLeu3-A(1-7) in a gel formulation — Gel will be applied to the wound once daily for four weeks (treatment period). Gel will have either no active ingredient (placebo), 0.03% or 0.01% active ingredient.
  Other Names: NorLeu3-Angiotensin(1-7); DSC127

SUMMARY:
The purpose of this study is to assess if the experimental drug, DSC127, is safe, how well it can be tolerated, and how different doses effect the healing of the chronic foot ulcers in diabetic subjects.

DETAILED DESCRIPTION:
This study is designed as a randomized, parallel-group, double-blind, placebo-controlled trial. After a 14-day baseline to evaluate ulcer healing to ensure DU are chronic, a 4-week active treatment followed by 8 weeks of observation and assessment of the treatment will compare the effects of two concentrations of DSC127 and placebo (n = 25 evaluable subjects per group; n=75 total evaluable subjects) to identify the optimal dose of DSC127. Sustained tissue integrity will be evaluated for all subjects during a follow-up period at study weeks 16 and 24.

Subjects will be randomized in a 1:1:1 ratio to one of the three treatment groups.

Group 1: Placebo Vehicle Control Group 2: 0.03% DSC127 in Vehicle Group 3: 0.01% DSC127 in Vehicle

The four week treatment period requires daily application of the treatment to the wound site. First application each week will be at the clinic and for the remainder of the week the patient self-administers the treatment.

If wound healing occurs during the treatment or assessment periods a final assessment visit is conducted and the integrity is assessed four and twelve weeks later (usually weeks 16 and 24 of the study).

ELIGIBILITY:
Inclusion Criteria:

* Have at least one chronic non-healing Wagner Grade 1 or Grade 2 plantar neuropathic diabetic ulcer between 1.0-6.0 cm2 on the midfoot or forefoot, including the toes but excluding the heel.
* ABI greater than 0.7 for neuroischemic or greater than 0.8 for neuropathic DU
* TcPO2 greater than 40 mm Hg or great toe systolic pressure greater than 50 mmHg
* Type I or Type II diabetes under metabolic control
* Female subjects must have a negative pregnancy test and be willing to use acceptable method of birth control for the duration of the study

Exclusion Criteria:

* Exposure to any investigational product within the last 30 days, or have known hypersensitivity to any of the study medication components
* Chronic renal insufficiency and/or chronic liver dysfunction
* Resting blood pressure (at the time of the initial visit of the Screening Period) which exceeds 160 systolic and/or 90 diastolic mmHg on 3 consecutive readings at least 15 minutes apart
* Malignancy of any kind
* Receiving hemodialysis or CAPD
* Current history of drug abuse, and/or known to be HIV positive
* Prior radiation therapy of the foot under study
* Current use of corticosteroids (within past 8 weeks), immunosuppressants (within past 8 weeks), or use of a biologic agent to include growth factors and skin equivalents (Regranex, Apligraft, or Dermagraft) in the past 90 days
* Ulcer is deemed clinically infected and requires topical antimicrobials or agents known to affect wound healing, or the subject has been taking systemic antibiotics for more than 7 days for any reason
* Sickle-cell anemia, Raynaud's or other peripheral vascular disease
* Wagner Grade 3 or higher DU, deep abscess or infection of the joint or tendon, or gangrene or osteomyelitis
* An EKG with a marked baseline prolongation of QT/QTc interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-10; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gere diZerega, MD, Study Director — US Biotest, Inc.
Locations (12):
- United States (12):
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Southern Arizona Limb Salvage Alliance (SALSA), Tucson, Arizona
  - Bay Area Footcare, Castro Valley, California
  - University of California, San Diego, San Diego, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - Passavant Area Hospital, Jacksonville, Illinois
  - Georgetown University Medical Center, Georgetown, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Eastern Carolina Foot & Ankle Specialists, Greenville, North Carolina
  - Warren General Hospital Wound Clinic, Warren, Pennsylvania
  - Renaissance Hospital Dallas, Dallas, Texas
  - Professional Education and Research Institute, Roanoke, Virginia

REFERENCES:
- [Background] Rodgers KE, Ellefson DD, Espinoza T, Roda N, Maldonado S, Dizerega GS. Effect of NorLeu3-A(1-7) on scar formation over time after full-thickness incision injury in the rat. Wound Repair Regen. 2005 May-Jun;13(3):309-17. doi: 10.1111/j.1067-1927.2005.130314.x. PMID 15953051
- [Background] Rodgers KE, Espinoza T, Felix J, Roda N, Maldonado S, diZerega G. Acceleration of healing, reduction of fibrotic scar, and normalization of tissue architecture by an angiotensin analogue, NorLeu3-A(1-7). Plast Reconstr Surg. 2003 Mar;111(3):1195-206. doi: 10.1097/01.PRS.0000047403.23105.66. PMID 12621191
- [Background] Rodgers K, Xiong S, Felix J, Roda N, Espinoza T, Maldonado S, Dizerega G. Development of angiotensin (1-7) as an agent to accelerate dermal repair. Wound Repair Regen. 2001 May-Jun;9(3):238-47. doi: 10.1046/j.1524-475x.2001.00238.x. PMID 11472620
- [Background] Rodgers KE, Roda N, Felix JE, Espinoza T, Maldonado S, diZerega G. Histological evaluation of the effects of angiotensin peptides on wound repair in diabetic mice. Exp Dermatol. 2003 Dec;12(6):784-90. doi: 10.1111/j.0906-6705.2003.00087.x. PMID 14714558
- [Result] Balingit PP, Armstrong DG, Reyzelman AM, Bolton L, Verco SJ, Rodgers KE, Nigh KA, diZerega GS. NorLeu3-A(1-7) stimulation of diabetic foot ulcer healing: results of a randomized, parallel-group, double-blind, placebo-controlled phase 2 clinical trial. Wound Repair Regen. 2012 Jul-Aug;20(4):482-90. doi: 10.1111/j.1524-475X.2012.00804.x. Epub 2012 Jun 7. PMID 22672145

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Vehicle Control: control placebo vehicle
- 0.03 % DSC127: 0.03% DSC127 in Vehicle Control
Period: Overall Study
Arm/Group | Placebo Vehicle Control | 0.03 % DSC127 | 0.01% DSC127
Started | 24 | 26 | 28
Completed | 24 | 26 | 27
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Vehicle Control | 0.03 % DSC127 | 0.01% DSC127 | Total
Number analyzed (Participants) | 24 | 26 | 28 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 21 | 24 | 62
  >=65 years | 7 | 5 | 4 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 56.8 (12.77) | 56.3 (10.35) | 53.1 (12.47) | 55.3 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 3 | 18
  Male | 16 | 19 | 25 | 60
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 28 | 78

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Parameter Will be the Proportion of Ulcers Healed by 12 Weeks as Defined as 100 % Epithelialized With no Drainage.
Time Frame: Healing to occur within 12 weeks of first treatment
Population: Intent-to-Treat Population
Measure: Number; unit: number of ulcers healed
Groups:
- Placebo: control placebo vehicle
- 0.03% DSC127: 0.03% DSC127 in Vehicle Control
Arm/Group | Placebo | 0.03% DSC127 | 0.01% DSC127
Number analyzed (Participants) | 24 | 26 | 27
number of ulcers healed | 8 [15.6 to 55.3] | 14 [33.4 to 73.4] | 8 [13.8 to 50.2]

2. Secondary Outcome: The Proportion of Subjects in Each Treatment Group Reporting Adverse Events.
Time Frame: Duration of subject's participation (24 weeks)
Population: Safety Population
Measure: Number; unit: patients
Arm/Group | Placebo Vehicle Control | 0.03 % DSC127 | 0.01% DSC127
Number analyzed (Participants) | 24 | 26 | 28
patients
  All Adverse Event | 23 | 26 | 28
  Serious Adverse Event | 5 | 4 | 4
  Related to Study Drug | 0 | 0 | 0

3. Secondary Outcome: The Rate of Re-epithelialization of the Ulcer Site.
Description: The overall healing rate of the ulcers, based on the percent of unhealed ulcer area re-epithelialized per week.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percent ulcer area re-epithelialized/wk
Arm/Group | Placebo | 0.03% DSC127 | 0.01% DSC127
Number analyzed (Participants) | 24 | 26 | 27
percent ulcer area re-epithelialized/wk | 10.5 (21.2) | 14.3 (12.8) | 9.0 (11.1)

4. Secondary Outcome: The Time to Re-epithelialization of the Ulcer Site.
Description: Average time to complete re-epithelialization of baseline ulcer area.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: Weeks
Arm/Group | Placebo Vehicle Control | 0.03 % DSC127 | 0.01% DSC127
Number analyzed (Participants) | 24 | 26 | 27
Weeks | 16.5 (1.77) | 12.4 (1.80) | 17.3 (1.53)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Maximum subject participation period.
Arm/Group | Placebo Vehicle Control | 0.03 % DSC127 | 0.01% DSC127
Serious Adverse Events (participants affected / at risk) | 5/24 | 4/26 | 4/28
Other Adverse Events (participants affected / at risk) | 16/24 | 15/26 | 18/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Vehicle Control (N=24) | 0.03 % DSC127 (N=26) | 0.01% DSC127 (N=28)
Acute Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Foot Amputation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Joint Arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Spinal Fusion Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Tendon Operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Vehicle Control (N=24) | 0.03 % DSC127 (N=26) | 0.01% DSC127 (N=28)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 2 (3)
Blood Glucose Increased (Investigations) | 1 (2) | 1 (1) | 2 (2)
Diabetic Foot (Metabolism and nutrition disorders) | 7 (10) | 7 (10) | 10 (22)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (3) | 5 (7)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 1 (1)
Skin Maceration (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (2)
Hypertension (Vascular disorders) | 1 (4) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor prepared an integrated clinical/statistical report. As this was a multicenter study, any publication/presentation of data was to include the entire study population. Publication/presentation of data from individual study centers is not allowed without explicit permission from US Biotest.